CLINICAL TRIAL: NCT06847776
Title: Longitudinal Evaluation of a Fracture Liaison Service
Acronym: FILFRA
Status: Enrolling by invitation | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Marine FAUNY, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2025PI010
Record Dates: First submitted 2025-02-07; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Osteoporosis
Keywords: osteoporosis; fractures; DXA; CT
MeSH Terms: conditions — Osteoporosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The major objective of this study is to evaluated osteoporosis prevalence, both on computed tomography (CT) and dual x ray absorptiometry (DXA) in patients included in a fracture liaison service (FLS).

The secondary objectives are to evaluate the prevalence of antiosteoporotic treatments indication, of new fractures or mortality; to identify the risk factor for osteoporosis; the study the treatment's observance; to identify the screening threshold to diagnose osteoporosis on CT.

ELIGIBILITY:
Inclusion Criteria:

* age >= 50 years
* Bone fracture due to a fall

Exclusion Criteria:

* patient's opposition

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients included in the fracture liaison service
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2030-01-02 (Estimated); Study Completion 2030-01-02 (Estimated)

PRIMARY OUTCOMES:
Osteoporosis prevalence on DXA and CT | during the evaluation in the fracture liaison service FLS and evry year until 5 years

SECONDARY OUTCOMES:
prevalnce of treatment for osteoporosis | during the evaluation in FLS and every year until 5 years
prevalence of new fractures at 1-3 and 5 years | during the evaluation in FLS and at 1, 3 and 5 years
identification of osteoporosis risk factors | at the inclusion in FLS
definition of the CT threshold for bone fragility in this population; | at the inclusion in FLS
study of the correlation dual x ray absorptiometry and computed tomography bone fragility evaluation | at the inclusion in FLS
study of the correlation between FRAX score and DXA | at the inclusion in FLS
study of the correlation between FRAX score and Trabecular bone score TBS | at the inclusion in FLS
study of the correlation between FRAX score and lean mass | at the inclusion in FLS

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided